CLINICAL TRIAL: NCT00631813
Title: A Double-Blind Placebo-Controlled Dose-Finding Trial to Evaluate the Efficacy and Safety of R093877 in Patients With Chronic Idiopathic Constipation
Brief Title: Efficacy and Safety Study of Prucalopride for the Treatment of Chronic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRU-INT-2
Record Dates: First submitted 2008-02-06; First posted 2008-03-10 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Prucalopride 0.5 mg
  Interventions: Drug: Prucalopride
- 2 (Active Comparator): Prucalopride 1 mg
  Interventions: Drug: Prucalopride
- 3 (Active Comparator): Prucalopride 2 mg
  Interventions: Drug: Prucalopride
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prucalopride — 0.5 mg bid
  Other Names: Resolor
  Arms: 1
Drug: Prucalopride — 1 mg bid
  Other Names: Resolor
  Arms: 2
Drug: Prucalopride — 2 mg bid
  Other Names: Resolor
  Arms: 3
Drug: Placebo — bid
  Arms: 4

SUMMARY:
The purpose of this study is to determine which dose of prucalopride is safe and effective in patients with chronic constipation.

Hypothesis:

Prucalopride 1 and 2 mg bid are safe and effective for the treatment of chronic constipation whereas 0,5 mg is a suboptimal dose.

DETAILED DESCRIPTION:
This is a phase II trial with a parallel-group design, consisting of a drug-free run-in phase (phase 1), followed by a placebo controlled double-blind phase (phase 2). Patients will receive either R093877 0.5 mg b.i.d., 1 mg b.i.d. or 2 mg b.i.d. or placebo for a period of 12 weeks.

Phase 1 is a run-in period of 4 weeks duration, during which the bowel habit is documented and the existence of constipation confirmed. At the start of this period all existing laxative medication is withdrawn and patients will be instructed not to change their dietary habits, in particular their fiber intake during the trial. Patients will enter the double-blind phase if constipation has been shown to be present during the run-in period.

If the definition of constipation was not met during the 4 weeks of the run-in period, the patient will be considered ineligible for the double-blind period.

Phase 2 is a double-blind, randomized, placebo-controlled phase, in which patients will be treated for 12 weeks with either 0.5 mg, 1 mg or 2 mg of R093877 or placebo given twice daily (one capsule is taken before breakfast and one is to be taken before the evening meal).

Patients admitted to the double blind treatment period will be randomly allocated to one of the 4 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-70 years;
2. History of constipation, i.e., the subject reported the occurrence of two or more of the following criteria for at least 6 months before the selection visit:

   * two or fewer spontaneous* bowel movements a week,
   * lumpy (scyballae) and/or hard stools at least ¼ of the stools,
   * sensation of incomplete evacuation after at least ¼ of the stools,
   * straining at defaecation at least ¼ of the time. *The above criteria were only applicable for spontaneous bowel movements i.e., not preceded within a 24-hour period by the intake of a laxative agent. Subjects who never had a spontaneous bowel movement were considered constipated and eligible to enter the double-blind phase of the trial.
3. Constipation being severe and causing disability; the subject's occupational, social and recreational activities were governed by his/her constipation and efforts to attain relief;
4. Normal inhibition pattern of the external anal sphincter during straining i.e., relaxation of the m.puborectalis and a distal displacement of the rectal canal (digital examination and/or electromyographic and/or manometric evidence was acceptable);
5. Poor results with routine laxative treatment and diet counselling;
6. Constipation of a functional, i.e., idiopathic nature;
7. Written or oral witnessed informed consent;
8. Availability for follow-up during the trial period.

Exclusion Criteria:

1. Constipation thought to be drug-induced;
2. Presence of secondary causes of constipation, i.e., subjects suffering from types or causes of constipation other than idiopathic constipation, for instance: endocrine disorders, metabolic disorders, or neurologic disorders;
3. Congenital megacolon/megarectum;
4. History of previous abdominal surgery (other than hysterectomy, surgery for Meckel's diverticle, appendectomy, cholecystectomy, inguinal hernia repair, splenectomy, nephrectomy or fundoplication) thought to be the primary cause of constipation;
5. Known or suspected organic disorders of the large bowel, i.e., obstruction, carcinoma or inflammatory bowel disease;
6. Active proctological conditions thought to be responsible for the constipation;
7. Presence of the following ECG abnormalities:

   * 2nd or 3rd degree of AV-block,
   * prolonged QT-times (> 460 ms),
   * bradycardia;
8. Use of concomitant medication that might cause QT-prolongation;
9. Use of diuretics not associated with potassium sparing effects;
10. Known illnesses or conditions such as severe cardiovascular or lung disease, neurologic or psychiatric disorders (including substance abused dependence but with the exception of nicotine), alcoholism, cancer or AIDS and other gastrointestinal or endocrine disorders;
11. Impaired renal function;
12. Presence of a serum amylase, a serum glutamic-oxaloacetic transaminase (SGOT) or a serum glutamic-pyruvic transaminase (SGPT) concentration of > 2 times the normal limit;
13. Presence of clinically significant abnormalities of blood chemistry, other than those mentioned under 9-10, haematology or urinalysis at selection;
14. Pregnancy or wish to become pregnant during the trial. ;
15. Breast-feeding;
16. Investigational drug received in the 30 days preceding the trial;
17. Inability or unwillingness to return for required follow-up visits;
18. Reliability and physical state preventing proper evaluation of a drug trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 1995-11; Primary Completion 1997-04 (Actual); Study Completion 1997-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy and to compare the effects of 0.5 mg, 1 mg or 2 mg of R093877 versus placebo | 12 weeks

SECONDARY OUTCOMES:
Evaluation of the effects of R093877 on symptoms associated with chronic constipation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: P. Van Eeghem, MD, Principal Investigator — Onze Lieve Vrouw Hospital

REFERENCES:
- [Derived] Emmanuel A, Cools M, Vandeplassche L, Kerstens R. Prucalopride improves bowel function and colonic transit time in patients with chronic constipation: an integrated analysis. Am J Gastroenterol. 2014 Jun;109(6):887-94. doi: 10.1038/ajg.2014.74. Epub 2014 Apr 15. PMID 24732867